CLINICAL TRIAL: NCT04328220
Title: Diagnostic Role of Chest Ultrasound in Children Presenting With Respiratory Distress in PICU Compared to Chest X-ray
Brief Title: Diagnostic Role of Chest Ultrasound in Children Presenting With Respiratory Distress in Pediatric Intensive Care Unit (PICU) Compared to Chest X-ray
Acronym: PICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Kotb, principlal investigator, Assiut University
Other Study IDs: chest US in PICU
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pediatric Respiratory Diseases
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: chest ultrasound — A point-of-care lung ultrasound exam will be performed within 24h of admission to PICU and serial follow up according to each case.
  chest x-ray will be performed for comparison with ultrasound findings.
  Other Names: Chest x-ray

SUMMARY:
The use of POCUS in pediatrics is gaining momentum, and whilst pediatric specific data remains limited when compared to adult critical care, there is growing pediatric evidence demonstrating the high sensitivity and specificity of lung POCUS in the diagnosis of pneumonia, bronchiolitis, pleural effusion and pneumothorax. the American Academy of Pediatrics policy statement cautions that "clinicians should be aware that point of care ultrasonography is better used as a rule in and not a rule out diagnostic modality".

DETAILED DESCRIPTION:
In recent years, the use of point-of-care ultrasound (PoCUS), understood as the bedside ultrasound examination of the patient by the physician in charge, has been increasing in paediatric patients for the investigation of pulmonary, pleural and diaphragmatic disease, following its use in adult patients, in whom the technique has been developing for more than a decade, and whose ultrasound semiotics can be safely extrapolated to the paediatric age group. The unossified costal cartilage and sternum and thinner adipose subcutaneous tissue in children provide ideal acoustic windows.

This study aims to compare the use of bedside lung US to portable chest X-ray regarding sensitivity, specificity, safety and accuracy in identifying the etiology of respiratory distress among children admitted to the PICU.

ELIGIBILITY:
Inclusion Criteria:

* Age >1month & <18years old
* All cases with clinically respiratory distress admitted in PICU Assiut University Children Hospital either connected to mechanical ventilation or not.

Exclusion Criteria:

1. Neonate.
2. Congenital anomalies of respiratory tract.
3. Cardiac diseases either congenital or acquired.
4. Traumatic patients.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — up to 18 Years
Study Population: Pediatric patients age 1 month and less than 18 years old with a clinical diagnosis of acute respiratory distress admitted in PICU Assiut University Children Hospital either connected to mechanical ventilation or not.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of point-of-care lung ultrasound examination in identifying the etiology of respiratory distress among patients admitted to the PICU. | baseline
  The sensitivity and specificity of the lung ultrasound in identifying the etiology of respiratory distress will be determined by comparison with bedside chest x ray.

REFERENCES:
- [Background] Quercia M, Panza R, Calderoni G, Di Mauro A, Laforgia N. Lung Ultrasound: A New Tool in the Management of Congenital Lung Malformation. Am J Perinatol. 2019 Jul;36(S 02):S99-S105. doi: 10.1055/s-0039-1692131. Epub 2019 Jun 25. PMID 31238368
- [Background] Supakul N, Karmazyn B. Ultrasound of the pediatric chest--the ins and outs. Semin Ultrasound CT MR. 2013 Jun;34(3):274-85. doi: 10.1053/j.sult.2012.12.001. PMID 23768893
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Bouhemad B, Zhang M, Lu Q, Rouby JJ. Clinical review: Bedside lung ultrasound in critical care practice. Crit Care. 2007;11(1):205. doi: 10.1186/cc5668. PMID 17316468
- [Background] Basile V, Di Mauro A, Scalini E, Comes P, Lofu I, Mostert M, Tafuri S, Manzionna MM. Lung ultrasound: a useful tool in diagnosis and management of bronchiolitis. BMC Pediatr. 2015 May 21;15:63. doi: 10.1186/s12887-015-0380-1. PMID 25993984